CLINICAL TRIAL: NCT02266745
Title: A Phase 1, Open-Label, Dose-Escalation Study Evaluating the Safety, Pharmacokinetics, and Clinical Effects of Intravenously Administered PT-112 Injection in Subjects With Advanced Solid Tumors and Subsequent Dose Expansion Cohorts
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Clinical Effects of Intravenously Administered PT-112 Injection in Subjects With Advanced Solid Tumors and Subsequent Dose Expansion Cohorts
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Promontory Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-112-101
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors; CRPC; mCRPC; Metastatic Castrate-resistant Prostate Cancer; PT-112; Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site
Keywords: PT-112
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site

STUDY DESIGN:
Intervention Model Description: Subjects enrolled in Cohort D Part 2 will be randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Arm 1: PT-112 injection (Experimental): Arm 1: PT-112 Injection, administered by intravenous infusion, biweekly 360 mg/m2
  Interventions: Drug: PT-112 Injection
- Arm 2: PT-112 injection (Experimental): Arm 2: PT-112 Injection, administered by intravenous infusion, biweekly 250 mg/m2
  Interventions: Drug: PT-112 Injection
- Arm 3: PT-112 injection (Experimental): Arm 3: PT-112 Injection, administered by intravenous infusion, 360 mg/m2 for two doses, 250 mg/m2 for subsequent doses
  Interventions: Drug: PT-112 Injection

INTERVENTIONS:
Drug: PT-112 Injection
  Other Names: PT-112

SUMMARY:
This is a Phase 1/2, open-label, multi-center, non-randomized, dose-escalation study to be conducted in two parts: the Dose Escalation Phase and the Dose Expansion Phase. The Dose Escalation Phase will determine the Maximum Tolerated Dose (MTD) and recommended Phase 2 dose(s) (RP2D) of PT-112 Injection and evaluate its safety and tolerability, and PK (pharmacokinetics).

The Dose Escalation Phase is complete and no longer enrolling.

The Dose Expansion Phase has two cohorts: one cohort for the study of PT-112 in patients with thymoma and thymic carcinoma (Cohort A), and one cohort for the study of PT-112 in metastatic castrate-resistant prostate cancer (mCRPC) (Cohort D).

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multi-center, non-randomized, dose-escalation study to be conducted in two parts: the Dose Escalation Phase, and the Dose Expansion Phase

The Dose Escalation Phase and the Dose Expansion Thymoma Cohort are complete and no longer enrolling.

The Dose Expansion Phase of the study of PT-112 in metastatic castrate-resistant prostate cancer (mCRPC) is open and enrolling.

ELIGIBILITY:
Key Inclusion Criteria:

* Male >/= 18 years of age
* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Document current evidence of metastatic castration-resistant prostate cancer (mCRPC), where metastatic status is defined as having documented metastatic lesion(s) on either bone scan or CT/MRI scan.
* Patients who have received at least three prior intended life-prolonging therapies for metastatic disease.
* Eastern Collaborative Oncology Group (ECOG) Performance Status of 0-1.
* Progressive disease, either measurable on physical examination or imaging by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or PCWG3 or by informative tumor marker(s).
* Adequate organ function based on laboratory values.
* If there is a known history of brain metastases, either treated or untreated, the disease must be stable.

Key Exclusion Criteria:

* Any cytotoxic chemotherapy within 21 days prior to initiation of study drug.
* Any immunomodulatory drug therapy, anti-neoplastic hormonal therapy, immunosuppressive therapy, corticosteroids, or growth factor treatment within 14 days prior to initiation of study drug.
* Bone marrow reserve which is not adequate for participation in this trial.
* Radiotherapy within 14 days prior to baseline.
* Fraction of radiotherapy to >25 % of active bone marrow.
* Major surgery within 28 days prior to initiation of study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2014-07; Primary Completion 2024-08-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Initial design: Comparison of two dose levels, administered on Days 1 and 15 of each 28-day cycle: | 28-day cycle
  [ ] Define the recommended dose level for PT-112 for pivotal studies based on the risk/benefit ratio across Arms 1, 2 and 3.
  Cohort D only
Modified design: Define the recommended dose and schedule for PT-112 for pivotal studies | 28-day cycle
  Define the recommended dose and schedule for PT-112 for pivotal studies.
  Cohort D only

SECONDARY OUTCOMES:
Disease Control Rate by disease manifestation, evaluated using PCWG3-modified RECIST criteria | up to 24 months
  Cohort D only
Objective Response Rate (ORR) in patients with RECIST-measurable disease, evaluated using PCWG3-modified RECIST criteria | up to 24 months
  Cohort D only
Median duration of response (DOR) as defined by PCWG3-modified RECIST criteria | up to 24 months
  Cohort D only
Percentage of patients achieving PSA50 as defined by PCWG3 criteria | up to 24 months
  Cohort D only
Percentage of patients who are CTC nonzero at baseline and with 0 CTCs/mL in one or more post-baseline samples (i.e., CTC0) | up to 24 months
  Cohort D only
Percentage of patients who have ≥ 3 CTCs at baseline and ≤ 3 CTCs in one or more post-baseline samples (i.e., CTC conversion) | up to 24 months
  Cohort D only
Median radiographic progression free survival (rPFS) by PCWG3 criteria | up to 24 months
  Cohort D only
Median overall survival (OS) | up to 24 months
  Cohort D only
Time to PSA progression by PCWG3 criteria | up to 24 months
  Cohort D only
Change in disease related pain based on ACS Daily Pain Diary assessment | up to 24 months
  Cohort D only

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D. Karp, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (25):
- United States (17):
  - Arizona, Phoenix, Arizona
  - Tucson, Tucson, Arizona
  - Duarte, Duarte, California
  - Colorado, Aurora, Colorado
  - Jacksonville, Jacksonville, Florida
  - Orlando, Orlando, Florida
  - Indianapolis, Indianapolis, Indiana
  - Boston, Boston, Massachusetts
  - Minneapolis, Minneapolis, Minnesota
  - Rochester, Rochester, Minnesota
  - Omaha, Omaha, Nebraska
  - Albuquerque, Albuquerque, New Mexico
  - Brooklyn, Brooklyn, New York
  - New York, New York, New York
  - Durham, Durham, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle, Seattle, Washington
- France (8):
  - Besançon, Besançon
  - Bordeaux, Bordeaux
  - Caen, Caen
  - Clermont-Ferrand, Clermont-Ferrand
  - Marseille, Marseille
  - Nice, Nice
  - Paris, Paris
  - Rennes, Rennes

REFERENCES:
- [Derived] Karp DD, Camidge DR, Infante JR, Ames TD, Price MR, Jimeno J, Bryce AH. Phase I study of PT-112, a novel pyrophosphate-platinum immunogenic cell death inducer, in advanced solid tumours. EClinicalMedicine. 2022 May 27;49:101430. doi: 10.1016/j.eclinm.2022.101430. eCollection 2022 Jul. PMID 35747193